CLINICAL TRIAL: NCT06370208
Title: Study to Investigate the Prophylactic Effect of Probiotic Streptococcus Salivarius eK12 Supplementation Against Recurrent Streptococcus Pyogenes (GAS) Bacterial Pharyngotonsillitis in Children: A Randomized, Double-blind Controlled Clinical Trial
Brief Title: Prophylactic Effect of Probiotic Streptococcus Salivarius eK12 Against Recurrent Streptococcus Pyogenes Pharyngotonsillitis Infection in Pediatrics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LUMHS/REC/-496/11.11.2024
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Streptococcus Pyogenes Pharyngotonsillitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic supplement group (Experimental): Participants in this group will receive probiotic Streptococcus salivarius eK12 (Bactoblis® EVOLcontaining ca. 1 billion CFU of Streptococcus salivarius eK12/capsule) as daily one capsule (to be slowly dissolved in the mouth before sleeping at night time) for 3-months. There will be a further 3-months follow-up period.
  Interventions: Dietary Supplement: Probiotic Bactoblis® EVOL (Streptococcus salivarius eK12)
- Control group (No Intervention): Participants in this group will not receive probiotic Streptococcus salivarius eK12 (Bactoblis® EVOL).

INTERVENTIONS:
Dietary Supplement: Probiotic Bactoblis® EVOL (Streptococcus salivarius eK12) — Bactoblis® EVOL: containing one billion CFU of probiotic Streptococcus salivarius eK12
  Arms: Probiotic supplement group

SUMMARY:
Recurrent Group A Streptococcus (GAS) infections, primarily presenting as strep throat, are a significant health concern in pediatric populations, leading to symptoms like sore throat, fever, and swollen lymph nodes. GAS is highly contagious and can spread easily among children in close-contact environments like schools and daycare centers, often resulting in frequent re-infections. Managing these recurrent infections typically requires antibiotics, but reliance on antibiotics carries risks, including resistance development, gut microbiota disruption, and various side effects. Probiotic therapy, particularly with Streptococcus salivarius K12, has shown promise as a preventive approach, utilizing competitive exclusion and antimicrobial production to inhibit GAS growth in the oral cavity. Recent studies have advanced this with the development of S. salivarius eK12, a re-engineered strain that enhances efficacy against GAS by preventing the survival-promoting interactions between the probiotic and pathogenic bacteria. This modified strain, now registered as Bactoblis® EVOL in Italy (EU), holds potential as an effective version to reduce the incidence and severity of GAS infections without the drawbacks of antibiotic therapy.

DETAILED DESCRIPTION:
The primary aim of this clinical trial is to evaluate whether prophylactic use of S. salivarius eK12 can effectively reduce the frequency and severity of strep throat episodes in children. By assessing the efficacy of S. salivarius eK12 supplementation, this study seeks to provide insights into its potential as a non-antibiotic preventive strategy for recurrent strep throat infections in pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-10 years.
* Recent history of documented recurrent episodes of Streptococcus pyogenes pharyngo- tonsillitis infection in the last 6 months, or 4 or more episodes in the last 12 months (S.

pyogenes infection being defined as: McIsaac score with clinical score ≥ 2 plus confirmation of S. pyogenes presence with rapid throat swab (RAD) method or McIsaac score =5.

* Willingness to comply with the study protocol and attend scheduled follow-up visits.
* Written informed consent obtained from the parent or legal guardian.

Exclusion Criteria:

* Children with known allergies or hypersensitivity to probiotics or any components of the study product.
* Current use of antibiotics or within the past 30 days.
* Used oral colonizing probiotics in the last 6 months.
* Presence of severe underlying medical conditions affecting the immune system or gastrointestinal tract.
* Participation in other clinical trials involving investigational drugs or interventions.
* Inability to adhere to the study requirements due to logistical or social reasons.
* History of rheumatic disorders, bronchospasm, severe asthma, or allergy requiring corticosteroids.
* Past tonsillectomy or an indication for adeno-tonsillectomy; or severe respiratory or systemic disorders
* Individuals immunocompromised or had a condition favouring recurrent Acute Otitis Media (AOM), including severe atopy, acquired or congenital immunodeficiency, cleft palate, craniofacial abnormalities, obstructive adenoids, a chronically ruptured eardrum, sleep apnoea, or tympanostomy tubes
* Children undergoing current pharmacological therapies to prevent recurrent respiratory infections.
* Any other medical condition or circumstance that, in the investigator's judgment, would compromise the safety of the participant or the integrity of the study.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Streptococcus pyogenes pharyngotonsillitis infection | 6-months
  Number of episodes of Streptococcus pyogenes pharyngotonsillitis infection
Probiotic safety and tolerability | 6-months
  Incidences of any side effects

SECONDARY OUTCOMES:
Protection against viral infection | 6-months
  Number of incidences of viral throat infection
Protection against Acute Otitis Media infection | 6-months
  Number of incidences of Acute Otitis Media infection
Protection against respiratory infection | 6-months
  Number of incidences of Tracheitis infection
Protection against Rhinitis | 6-months
  Number of incidences of Rhinitis
Protection against flu | 6-months
  Number of incidences of flu
Protection against Enteritis | 6-months
  Number of incidences of Enteritis infection
Protection against Stomatitis | 6-months
  Number of incidences of Stomatitis infection

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat University of Medical and Health Sciences, Jamshoro, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Pierro F, Veeraraghavan G, Kalaiselvan K, Ashif B, Jeyakumar L, Gopalakrishnan G, Cazzaniga M, Bertuccioli A, Tanda ML, Zerbinati N, Ujjan I, Bugti AA, Bano A, Gull Y, Mumtaz N, Khan A. In Vitro and In Vivo Safety Evaluation of Streptococcus salivarius eK12, a Genetically Modified Dietary Probiotic Derived from the Oral Probiotic S. salivarius K12. J Microbiol Biotechnol. 2025 Dec 9;35:e2509016. doi: 10.4014/jmb.2509.09016. PMID 41391486
- [Background] Di Pierro F, Bugti AA, Bano A, Kara M, Ujjan I, Mumtaz N, Gull Y, Cazzaniga M, Bertuccioli A, Tanda ML, Zerbinati N, Hameed S, Khan A. Study to evaluate the safety and tolerability of Streptococcus salivarius eK12, a genetically modified strain derived from the oral probiotic S. salivarius K12: Results from a randomized, double-blind, placebo-controlled, parallel-group clinical trial. Front Nutr. 2025 Dec 8;12:1701611. doi: 10.3389/fnut.2025.1701611. eCollection 2025. PMID 41438195
- [Result] Di Pierro F, Colombo M, Giuliani MG, Danza ML, Basile I, Bollani T, Conti AM, Zanvit A, Rottoli AS. Effect of administration of Streptococcus salivarius K12 on the occurrence of streptococcal pharyngo-tonsillitis, scarlet fever and acute otitis media in 3 years old children. Eur Rev Med Pharmacol Sci. 2016 Nov;20(21):4601-4606. PMID 27874935
- [Result] Di Pierro F, Colombo M, Zanvit A, Rottoli AS. Positive clinical outcomes derived from using Streptococcus salivarius K12 to prevent streptococcal pharyngotonsillitis in children: a pilot investigation. Drug Healthc Patient Saf. 2016 Nov 21;8:77-81. doi: 10.2147/DHPS.S117214. eCollection 2016. PMID 27920580
- [Result] Di Pierro F, Colombo M, Zanvit A, Risso P, Rottoli AS. Use of Streptococcus salivarius K12 in the prevention of streptococcal and viral pharyngotonsillitis in children. Drug Healthc Patient Saf. 2014 Feb 13;6:15-20. doi: 10.2147/DHPS.S59665. eCollection 2014. PMID 24600248
- [Result] Di Pierro F, Donato G, Fomia F, Adami T, Careddu D, Cassandro C, Albera R. Preliminary pediatric clinical evaluation of the oral probiotic Streptococcus salivarius K12 in preventing recurrent pharyngitis and/or tonsillitis caused by Streptococcus pyogenes and recurrent acute otitis media. Int J Gen Med. 2012;5:991-7. doi: 10.2147/IJGM.S38859. Epub 2012 Nov 30. PMID 23233809
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23231486/